CLINICAL TRIAL: NCT06147596
Title: Heading in Football: Impact on Neural Blood Biomarkers
Acronym: HEADLINE
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Koninklijke Nederlandse VoetbalBond (KNVB) (Unknown)
Responsible Party: Principal Investigator, Prof. dr. Jaap Oosterlaan, Director Follow me programme, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL83396.018.23
Record Dates: First submitted 2023-10-05; First posted 2023-11-27 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-01

CONDITIONS: Head Injury, Minor; Concussion, Mild; CTE - Chronic Traumatic Encephalopathy; Neurodegeneration
Keywords: Heading; Soccer; Head impact; Blood biomarker; Neurodegeneration
MeSH Terms: conditions — Craniocerebral Trauma; Brain Concussion; Chronic Traumatic Encephalopathy; Nerve Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood is collected with the possibility of DNA analysis in the future.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Soccer: Healthy volunteers that participate in the study by playing a regular soccer game for the sake of the HEADLINE study
  Interventions: Other: Head impact exposure

INTERVENTIONS:
Other: Head impact exposure — The cohort is exposed to naturalistic head impacts (heading) during voluntary participation in a soccer match. All participants are regular soccer players and are therefore not exposed to excessive head impacts compared to their regular exposure.

SUMMARY:
The goal of this observational study is to evaluate the safety of heading in football. We will study the release of biomarkers in blood that reflect microscopic neural damage. The main questions this study aims to answer are:

* Does participation in a football match lead to a change in biomarkers that reflect microscopic neural damage?
* Is the dose of exposure during a football match related to the magnitude of change in biomarkers that reflect microscopic neural damage?

Participants will participate in a regular football match and provide blood samples before and right after the football match. The football match will be recorded on video to count the number of headers of all participants.

DETAILED DESCRIPTION:
The objective of this prospective observational study is to determine the potential impact of ball heading in football on brain integrity as assessed by blood biomarkers for neural damage in a real-world setting. Healthy amateur football players will be recruited to participate in the study. Participants will be invited to play a regular football match for investigation purposes. They will provide a blood sample within one hour before the start of the match and a second blood sample within one hour after the match. Participants will be asked to provide a third blood sample within 48 hours after participation, but this is not obligatory. The football match will be recorded on video to determine the number of head impacts of all participants. Furthermore, participants will wear heart rate sensors and local positioning sensors to determine the internal and external training load and account for the possible confounding effects of exercise on neural blood biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Member of the KNVB;
* 18 years or older;
* Male
* Self-reported fitness to play 70-90 minutes (absence of injury).

Exclusion Criteria:

* Sustained a head injury in the last year;
* History or current neurological condition;
* Regular participation in other contact sports (e.g. rugby, American football, ice hockey, fighting sports);
* (Former) military personnel with a history of fighting/blast exposure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All senior amateur football players will be invited to participate in the study. An amateur population is chosen because of the great number of participants and the resulting societal relevance of the research question.
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Concentration of serum neurofilament light protein | T0 (<1hour pre-match), T1 (<1hour post-match), T2 (<48hour post-match)
  The difference in serum neurofilament light protein between pre-match samples and post-match samples.

SECONDARY OUTCOMES:
Concentration of serum S100B protein | T0 (<1hour pre-match), T1 (<1hour post-match), T2 (<48hour post-match)
  The difference in serum S100B protein between pre-match samples and post-match samples.
Concentration of serum p-tau protein | T0 (<1hour pre-match), T1 (<1hour post-match), T2 (<48hour post-match)
  The difference in serum p-tau protein between pre-match samples and post-match samples.
Concentration of serum Neuron Specific Enolase protein | T0 (<1hour pre-match), T1 (<1hour post-match), T2 (<48hour post-match)
  The difference in serum Neuron Specific Enolase protein between pre-match samples and post-match samples.
Concentration of serum Glial Fibrillary Acidic Protein | T0 (<1hour pre-match), T1 (<1hour post-match), T2 (<48hour post-match)
  The difference in serum Glial Fibrillary Acidic Protein between pre-match samples and post-match samples.
Concentration of serum beta-synuclein | T0 (<1hour pre-match), T1 (<1hour post-match), T2 (<48hour post-match)
  The difference in serum beta-synuclein between pre-match samples and post-match samples.

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Oosterlaan, Prof.Dr., Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
We intend to make IPD available to other researchers. However, we still need to develop the plan in collaboration with the privacy officer and legal research support.